CLINICAL TRIAL: NCT03705234
Title: HPS-4/TIMI 65/ORION-4: A Double-blind Randomized Placebo-controlled Trial Assessing the Effects of Inclisiran on Clinical Outcomes Among People With Atherosclerotic Cardiovascular Disease
Brief Title: A Randomized Trial Assessing the Effects of Inclisiran on Clinical Outcomes Among People With Cardiovascular Disease
Acronym: ORION-4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: The TIMI Study Group (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTSU_MDCO_PCS-17-01
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Inclisiran; PCSK9; Cardiovascular; LDL Cholesterol; Cholesterol; Lipid; RNA interference
MeSH Terms: conditions — Atherosclerosis | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Inclisiran sodium 300 milligrams (mg) will be administered as a SC injection at randomization, 3 months and then every 6 months.
  Interventions: Drug: Inclisiran
- Placebo (Placebo Comparator): Placebo will be administered as SC injections of saline solution at randomization, 3 months and then every 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran — Inclisiran is a small interfering ribonucleic acid (RNA) that inhibits PCSK9 synthesis.
  Arms: Inclisiran
Drug: Placebo — Placebo will be supplied as sterile normal saline (0.9% sodium chloride in water for injection).
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
ORION-4 is a research study coordinated by the University of Oxford and co-sponsored by The University of Oxford and Novartis (Protocol: CTSU_MDCO-PCS-17-01 (CKJX839B12301)). The study aims to find out if a new cholesterol-lowering injection (inclisiran) safely lowers the risk of heart attacks and strokes in people who have already had one of these conditions, or who have had an operation or procedure to treat blocked arteries.

DETAILED DESCRIPTION:
The ORION-4 study aims to provide evidence about both the efficacy and safety of inclisiran. Inclisiran is a PCKS9 synthesis inhibitor which has been found to reduce LDL-cholesterol by about 50-60%. ORION-4 will investigate the effects of inclisiran on major adverse cardiovascular events.

The study is intended to be conducted at approximately 180 clinical sites in the UK and the USA. Approximately 15,000 participants aged 40 years or older for men, and 55 years or older for women, with pre-existing atherosclerotic cardiovascular disease will be randomized between inclisiran sodium 300 mg and matching placebo (given by subcutaneous injection on the day of randomization, at 3 months and then every 6-months) in a 1:1 ratio for a planned median duration of about 5 years.

ELIGIBILITY:
Inclusion Criteria

History or evidence of at least one of the following:

* Prior MI; or
* Prior ischemic stroke; or
* Peripheral artery disease as evident by prior lower extremity artery revascularization or aortic aneurysm repair.

Minimum age is 40 years for men and 55 years for women

Exclusion Criteria

None of the following must be satisfied (based on self-reported medical history):

* Acute coronary syndrome or stroke less than 4 weeks before the Screening visit or during the Run-in period;
* Coronary revascularization procedure planned within the next 6 months;
* Known chronic liver disease;
* Current or planned renal dialysis or transplantation;
* Previous exposure to inclisiran or participation in a randomized trial of inclisiran;
* Previous (within about 3 months), current or planned treatment with a monoclonal antibody targeting PCSK9, or with a drug known to be contra-indicated with inclisiran (none currently known);
* Known to be poorly compliant with clinic visits or prescribed medication;
* Medical history that might limit the individual's ability to take trial treatments for the duration of the study (e.g. severe respiratory disease; cancer or evidence of spread within approximately the last 5 years, other than non-melanoma skin cancer; or history of alcohol or substance misuse) or may put the individual at significant risk in the opinion of the investigator (or their authorised deputy) if he/she were to participate in the trial;
* Women of child-bearing potential, current pregnancy, or lactation;
* Current participation in a clinical trial with an unlicensed drug or device; or
* Staff personnel directly involved with the study and any family member of the investigational study staff.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16124 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2049-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a major adverse cardiovascular event (MACE) | Median follow-up of 5-years
  Defined as time to first occurrence - during the scheduled treatment period - of:
  * Coronary heart disease (CHD) death;
  * Myocardial infarction;
  * Fatal or non-fatal ischemic stroke; or
  * Urgent coronary revascularization procedure.

SECONDARY OUTCOMES:
Number of participants with MACE among those recorded to be taking high-intensity statin at baseline | Median follow-up of 5-years
Number of participants with a composite of CHD death or myocardial infarction | Median follow-up of 5-years
Number of participants with cardiovascular death | Median follow-up of 5-years

CONTACTS AND LOCATIONS:
Overall Officials: Louise Bowman, Principal Investigator — University of Oxford; Marion Mafham, Principal Investigator — University of Oxford; David Preiss, Principal Investigator — University of Oxford; Martin Landray, Principal Investigator — University of Oxford
Locations (2):
- TIMI Study Group, Boston, Massachusetts, United States
- CTSU, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Proposals for substudies must be approved by the Steering Committee. Procedure for accessing the data for this study are available on https://www.ndph.ox.ac.uk/data-access
Supporting Information: Study Protocol, SAP
Time Frame: After the main study results have been announced and published
Access Criteria: See URL
URL: https://www.ndph.ox.ac.uk/data-access

REFERENCES:
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512
- See also: Study website — https://www.orion4trial.org